CLINICAL TRIAL: NCT01753050
Title: A Quality Improvement Project for Goal-directed Intraoperative Hemodynamic Optimization in Patients Redo Hip Surgery
Brief Title: HIP Surgery - Hemodynamic Optimization Project
Acronym: HipHop
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, Sascha Treskatsch, Dr., Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HipHop; EA1/315/12 (Other: ethics commitee)
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Redo Hip Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (No Intervention): No specific hemodynamic optimization measures
- Hemodynamic optimization (Experimental): Hemodynamic optimization by stroke volume monitoring
  Interventions: Device: Stroke volume monitoring

INTERVENTIONS:
Device: Stroke volume monitoring — Pulse contour stroke volume monitoring
  Arms: Hemodynamic optimization

SUMMARY:
Several studies have demonstrated that goal-directed fluid therapy during high- risk-surgery reduces morbidity and length of hospital stay. This quality improvement is design to evaluate the implementation of an intraoperative goal-directed therapy, using a pulse contour analysis monitor to optimize the stroke volume, in patients undergoing redo-hip-surgery. The primary combined endpoints will be the incidence of postoperative complications and the secondary endpoints will be the decrease of hospital length of stay, length of ICU stay and hospital postoperative mortality. We amended another 130 patients getting crystalloid fluids in the hemodynamic optimization protocol.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing redo hip surgery
* age above 18 years
* signed informed consent

Exclusion Criteria:

* urgent or emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2012-12; Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
postoperative complications | 30days

SECONDARY OUTCOMES:
length of hospital and ICU stay | 30days

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Treskatsch, MD, Principal Investigator — Department of Anesthesiology and Operative Intensive Care Medicine, CCM and CVK
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine Campus Charité Mitte / Campus Virchow-Klinikum, Berlin, Germany

REFERENCES:
- [Derived] Trauzeddel RF, Leitner M, Dehe L, Nordine M, Piper SK, Habicher M, Sander M, Perka C, Treskatsch S. Goal-directed fluid therapy using uncalibrated pulse contour analysis and balanced crystalloid solutions during hip revision arthroplasty: a quality implementation project. J Orthop Surg Res. 2023 Apr 6;18(1):281. doi: 10.1186/s13018-023-03738-0. PMID 37024966
- [Derived] Habicher M, Balzer F, Mezger V, Niclas J, Muller M, Perka C, Kramer M, Sander M. Implementation of goal-directed fluid therapy during hip revision arthroplasty: a matched cohort study. Perioper Med (Lond). 2016 Dec 13;5:31. doi: 10.1186/s13741-016-0056-x. eCollection 2016. PMID 27999663